CLINICAL TRIAL: NCT05744934
Title: Interstage Monitoring Using an Implantable Loop Recorder: A Pilot Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Audrey Dionne, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-P00044387
Record Dates: First submitted 2023-02-03; First posted 2023-02-27 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Univentricular Heart
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: LUX-Dx™ — Placement of LUX-Dx at the time of stage 1 palliation

SUMMARY:
The primary objective of this investigation is to evaluate the feasibility and safety of implantable loop recorder implantation (using the LUX-DX™) in newborns undergoing stage 1 palliation. The secondary objective of the investigation is to evaluate the feasibility of continuous measurement of heart rate and arrhythmia using an implantable loop recorder (LUX-Dx™) during the interstage period.

An implantable loop recorder will be placed at the time of chest closure following stage 1 palliation (either at the time of index surgery or delayed). The device will be placed in a subclavicular pouch through the existing sternotomy incision. Participants will be in the study for 6 months to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single ventricle physiology undergoing stage 1 palliation in the 1st month of life

Exclusion Criteria:

* Prematurity (<36 weeks gestational age)
* Birth weight <2.5 kg
* Hybrid stage 1 palliation (patent ductus arteriosus stenting, bilateral pulmonary artery bands)
* Presence and/or need for devices sensitive to magnetic fields such as hearing aids, pacemaker, and other implanted devices.
* Clinical team does not think that the patient is a good candidate

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful ILR implantation at the time of surgery | At the time of stage 1 surgery, typically the first week of life
  Feasibility of ILR implantation
Number of patients with ILR related complication (any of: infection, erosion, device migration, foreign body rejection phenomena, formation of hematomas or seromas, local tissue reaction and/or tissue damage | Between the stage 1 and stage 2 surgery, typically until 4-6 months of age
  Safety of ILR implantation

SECONDARY OUTCOMES:
Number of patient who completed >70% planned ILR transmissions | Between the stage 1 and stage 2 surgery, typically until 4-6 months of age
Number of patients with arrhythmias | Between the stage 1 and stage 2 surgery, typically until 4-6 months of age
  Any arrhythmia, including supraventricular tachycardia, junctional ectopic tachycardia, ventricular tachycardia, atrioventricular block, pause >2.5 seconds
Number of patients with interstage complication | Between the stage 1 and stage 2 surgery, typically until 4-6 months of age
  Any complication, including unplanned emergency department visit, unscheduled hospital admission, unscheduled intensive care unit admission, arrhythmias, major interstage intervention, minor interstage intervention, cardiac arrest, death
Complications at the time of ILR removal | At stage 2 or 3 palliation, typically between 4 months and 4 years of age
  Defined as easily removed, removed with difficulty, removed with complication

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No